CLINICAL TRIAL: NCT07256769
Title: Synergic Role of Vitamin k, D-chiro Inositol and α-lactalbumin in Bone Homeostasis in Breast Cancer Patients Treated With Aromatase Inhibitors
Brief Title: Vitamin k, D-chiro Inositol and α-lactalbumin in Bone Homeostasis
Acronym: Synostea
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Marialuisa Appetecchia, Professor, Regina Elena Cancer Institute
Other Study IDs: RS 328/IRE/25
Record Dates: First submitted 2025-11-18; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis Secondary; Breast Cancer Females
Keywords: Vitamin K; d-chiro-inositol; α-lactalbumin; calcium; cancer treatment induced bone loss; vitamin d; synostea
MeSH Terms: interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Standard therapy
  Interventions: Dietary Supplement: Group 1: calcium carbonate/cholecalciferol
- Group 2: Synostea®
  Interventions: Dietary Supplement: Group 2: Synostea® (calcium carbonate/cholecalciferol/vitamin K/α-lactalbumin/ d-chiro-inositol)

INTERVENTIONS:
Dietary Supplement: Group 1: calcium carbonate/cholecalciferol — Intake of calcium carbonate 500 mg + cholecalciferol 2000 IU
  Groups: Group 1
Dietary Supplement: Group 2: Synostea® (calcium carbonate/cholecalciferol/vitamin K/α-lactalbumin/ d-chiro-inositol) — Intake of Synostea® : calcium carbonate 400 mg + cholecalciferol 2000 IU + vitamin K (menaquinone 50 μg) + α-lactalbumin (30 mg) + d-chiro-inositol (150 mg)
  Groups: Group 2

SUMMARY:
In women with breast cancer undergoing adjuvant hormone therapy, the marked tissue hypoestrogenism induced by therapy with aromatase inhibitors and/or tamoxifen ± GnRH analogues causes a significant acceleration in bone mass loss, with a consequent increased risk of fracture from the first year of therapy. It is therefore essential to start treatment with antiresorptive drugs and calcium and vitamin D supplementation. It has been hypothesized that vitamin K and α-lactalbumin have an effect in improving the absorption of calcium and vitamin D. In addition, vitamin K promotes gamma-carboxylation of osteocalcin, causing its activation and leading to increased incorporation of hydroxyapatite into the bone, resulting in increased calcium uptake from the blood and other tissues. Studies have reported that a combination of alendronate and vitamin K2 can lead to a decrease in the ratio of uncarboxylated osteocalcin to carboxylated osteocalcin, contributing to an increase in BMD, especially in the femoral neck. α-lactalbumin is able to increase the bioaccessibility of calcium due to its ability to prevent its precipitation at the neutral pH present in the absorptive tracts of the small intestine. Furthermore, α- lactalbumin has a binding site for vitamin D3, and the complexes formed by monomers of this protein and vitamin D have shown good stability in the presence of high vitamin concentrations. Inositol is a carbohydrate structurally similar to glucose which, in its isomeric form D-chiro-inositol, acts on bone remodeling by blocking the activation of osteoclasts through inhibition of the binding of RANK-L to its receptor present on pre-osteoclasts. Our hypothesis is that the use of the combination of vitamin K, α- lactalbumin, and D-chiro-inositol should improve the intestinal absorption of calcium and vitamin D, increasing the percentage of patients able to normalize serum levels of vitamin D and urinary calcium excretion (as a parameter of adequate calcium intake). This aspect, together with the direct effect of these components on bone remodeling, could enhance the anti-resorptive effect of standard therapy with bisphosphonates, improving the quantitative and qualitative parameters of bone. Therefore, we design a prospective randomized pilot study to assess efficacy of the combination of vitamin K, α-lactalbumin, and D-chiro-inositol, comparing patients with standard therapy and patients treated with Synostea®

DETAILED DESCRIPTION:
Recommendations regarding the ideal daily intake of calcium and vitamin D vary based on the anthropometric characteristics and comorbidities of patients. An adequate level of these two nutrients is recommended especially in patients undergoing treatment with anti-resorptive drugs used for both preventive and therapeutic purposes in osteoporosis. This occurs in women with breast cancer, in whom the marked tissue hypoestrogenism induced by adjuvant therapy (aromatase inhibitors and/or tamoxifen ± GnRH analogues) causes a significant acceleration in bone loss (CTIBL-Cancer Treatment-Induced Bone Loss), with a consequent increased risk of fracture from the first year of therapy. It is therefore essential to start treatment with antiresorptive drugs and calcium and vitamin D supplementation in order to safeguard bone health and prevent secondary osteoporosis.

Optimal serum concentrations of calcium and vitamin D play a central role in bone health, but insufficient intake can depend on numerous factors, including diet and the presence of other nutrients, as well as the body's ability to absorb them effectively. It has been hypothesized that vitamin K and α-lactalbumin improve the absorption of calcium and vitamin D. Vitamin K is a fat-soluble vitamin that comes in various forms, including vitamin K2 (menaquinone), which is involved in bone remodeling. It promotes gamma-carboxylation of osteocalcin, causing its activation and leading to increased incorporation of hydroxyapatite into bone, resulting in increased uptake of calcium from the blood and other tissues. High levels of the uncarboxylated form of osteocalcin, which is found in cases of vitamin K deficiency, have been associated with an increased risk of fractures despite adequate therapy with oral bisphosphonates. Studies have reported that a combination of alendronate and vitamin K2 can lead to a decrease in the ratio of uncarboxylated osteocalcin to carboxylated osteocalcin, contributing to an increase in BMD, especially in the femoral neck, thus reducing the risk of fragility fractures. α-Lactalbumin is a small acidic protein that has a binding site with high affinity for Ca++. The bioaccessibility of Ca++, i.e., the amount of micronutrient potentially available for absorption in the human body, depends on the amount of soluble calcium released from food processing during digestion. It has been hypothesized that binding to peptides such as α-lactalbumin may increase bioaccessibility due to its ability to prevent precipitation at the neutral pH present in the absorptive tracts of the small intestine. In addition, α-lactalbumin has a binding site for vitamin D3, and complexes consisting of monomers of this protein and vitamin D have shown good stability in the presence of high vitamin concentrations. It is also known from in vitro studies that α-lactalbumin can improve the intestinal absorption of D-chiro-inositol by as much as 10 times compared to the absence of this protein in the intestine.

The combination of vitamin K, α-lactalbumin, and D-chiro-inositol should improve the intestinal absorption of calcium and vitamin D, increasing the percentage of patients able to achieve normalization of serum vitamin D levels and urinary calcium excretion (understood as a parameter of adequate calcium intake). This aspect, together with the direct effect of these components on bone remodeling, could enhance the antiresorptive effect of standard bisphosphonate therapy, improving the quantitative and qualitative parameters of bone.

Inositol is a carbohydrate structurally similar to glucose which, in its D-chiro-inositol isomeric form, acts on bone remodeling by blocking the activation of osteoclasts through inhibition of the binding of RANK-L to its receptor present on pre-osteoclasts.

Therefore, we design a prospective randomized pilot study aims to evaluate the effect of synergistic effect of vitamin K, α-lactalbumin and D-chiro-inositol supplementation compared to standard therapy with calcium carbonate and vitamin D alone on calcium-phosphorus metabolism parameters and bone mineral density in patients with breast cancer treated with alendronate for the prevention of bone damage from hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* caucasian women aged between 35 and 70;
* diagnosed with breast cancer undergoing treatment with aromatase inhibitors or tamoxifen + GnRH analogues or aromatase inhibitors + GnRH analogues not started more than 12 months ago, about to start treatment with oral bone resorption inhibitors (alendronate);
* vitamin D levels below 30 ng/ml (test carried out no more than 6 months prior to the baseline/T0 visit)
* patients able to comply with the procedures and/or requirements of the study
* informed consent to participate in the study and data processing, written personally and/or through a witness, before any study-specific procedure is carried out

Exclusion Criteria:

* uncontrolled diabetes mellitus (HbA1c 8%), severe CRF (eGFR<30 ml/min);
* patients with primary or secondary hyperparathyroidism due to CRF;
* baseline vitamin D levels greater than 30 ng/ml;
* patients already being treated with anti-resorptive drugs;
* patients undergoing steroid therapy;
* patients undergoing treatment with other forms of vitamin D (calcifediol, calcitriol) or who require high doses of calcium (hypoparathyroidism);
* patients undergoing treatment with drugs that can affect calcium excretion (diuretics);
* inability to comply with the procedures required by the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women (aged between 35 and 70) with breast cancer undergoing treatment with aromatase inhibitors or tamoxifen + GnRH analogues or aromatase inhibitors + GnRH analogues, and about to start treatment with oral bone resorption inhibitors (alendronate), and meeting the other criteria
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of differences in mean vitamin D levels after six months in patients treated with calcium carbonate + cholecalciferoland patients treated with calcium carbonate + cholecalciferol + vitamin K + α-lactalbumin + d-chiro-inositol | 6 months
  Change in mean vitamin D levels in the two treatment groups after 6 months of therapy

SECONDARY OUTCOMES:
Evaluation of the differences in Hip Bone Mineral Density by D-XA between groups | 12 months
  To evaluate difference in the change from baseline in hip BMD (Bone Mineral Density) by dual x ray absorptiometry after 12 months between the 2 groups (standard vitamin d and calcium supplementation vs Synostea®)
Evaluation of the differences in lumbar fragility score by Radiofrequency Echographic Multi Spectrometry between groups | 12 months
  To evaluate difference in the change from baseline in lumbar fragility score by Radiofrequency Echographic Multi Spectrometry after 12 months between the 2 groups (standard vitamin d and calcium supplementation vs Synostea®)
Evaluation of the differences in serum levels of total calcium betweeeng groups after 12 months | 12 months
  To compare the changes in serum levels of total calcium after 12 months of treatment in the two groups (standard supplementationm with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of parathyroid hormone betweeen groups after 12 months | 12 months
  To compare the changes in serum levels of total calcium after 12 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of bone alkaline phosphatase betweeen groups after 12 months | 12 months
  To compare the changes in serum levels of bone alkaline phosphatase after 12 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of C-terminal telopeptide of type I collagen betweeen groups after 12 months | 12 months
  To compare the changes in serum levels of C-terminal telopeptide of type I collagen (CTX) after 12 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in 24-hour calciuria levels betweeen groups after 12 months | 12 months
  To compare the changes in 24-hour calciuria levels after 12 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of total calcium betweeen groups after 6 months | 6 months
  To compare the changes in serum levels of total calcium after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of parathyroid hormone betweeen groups after 6 months | 6 months
  To compare the changes in serum levels of parathyroid hormone after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of bone alkaline phosphatase betweeen groups after 6 months | 6 months
  To compare the changes in serum levels of bone alkaline phosphatase after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of C-terminal telopeptide of type I collagen betweeen groups after 6 months | 6 months
  To compare the changes in serum levels of C-terminal telopeptide of type I collagen (CTX) after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in 24-hour calciuria levels betweeen groups after 6 months | 6 months
  To compare the changes in 24-hour calciuria levels after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in Lumbar Bone Mineral Density by D-XA between groups | 12 months
  To evaluate difference in the change from baseline in lumbar BMD (Bone Mineral Density) by dual x ray absorptiometry after 12 months between the 2 groups (standard vitamin d and calcium supplementation vs Synostea®)
Evaluation of the differences in hip fragility score by Radiofrequency Echographic Multi Spectrometry between groups | 12 months
  To evaluate difference in the change from baseline in hip fragility score by Radiofrequency Echographic Multi Spectrometry after 12 months between the 2 groups (standard vitamin d and calcium supplementation vs Synostea®)
Evaluation of the differences in serum levels of total alkaline phosphatase betweeen groups after 6 months | 6 months
  To compare the changes in serum levels of total alkaline phosphatase after 6 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in serum levels of total alkaline phosphatase betweeen groups after 12 months | 12 months
  To compare the changes in serum levels of total alkaline phosphatase after 12 months of treatment in the two groups (standard supplementation with calcium and vitamin d vs Synostea®)
Evaluation of the differences in treatment adherence betweeen groups after 12 months | 12 months
  To assess the difference in treatment adherence between the two groups (standard supplementation with calcium and vitamin d vs Synostea®), evaluated using questionnaires created specifically for the study after 12 months.
Evaluation of the differences in treatment adherence betweeen groups after 6 months | 6 months
  To assess the difference in treatment adherence between the two groups (standard supplementation with calcium and vitamin d vs Synostea®), evaluated using questionnaires created specifically for the study after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Appetecchia, MD, Principal Investigator — Regina Elena National Cancer Insitute
Locations (2):
- Italy (2):
  - Santa Maria Goretti Hospital, Latina, Italy
  - Regina Elena National Cancer Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be published in GARRbox
Time Frame: Data will be available after study publication
Access Criteria: Data will be available for free
URL: https://gbox.garr.it/it/

REFERENCES:
- [Background] Atieh O, Daher J, Durieux JC, Abboud M, Labbato D, Baissary J, Koberssy Z, Ailstock K, Cummings M, Funderburg NT, McComsey GA. Vitamins K2 and D3 Improve Long COVID, Fungal Translocation, and Inflammation: Randomized Controlled Trial. Nutrients. 2025 Jan 16;17(2):304. doi: 10.3390/nu17020304. PMID 39861434
- [Background] Weaver CM. How sound is the science behind the dietary recommendations for dairy? Am J Clin Nutr. 2014 May;99(5 Suppl):1217S-22S. doi: 10.3945/ajcn.113.073007. Epub 2014 Mar 19. PMID 24646824
- [Background] Caputo M, Bona E, Leone I, Sama MT, Nuzzo A, Ferrero A, Aimaretti G, Marzullo P, Prodam F. Inositols and metabolic disorders: From farm to bedside. J Tradit Complement Med. 2020 Mar 24;10(3):252-259. doi: 10.1016/j.jtcme.2020.03.005. eCollection 2020 May. PMID 32670820
- [Background] Ranaldi G, Ferruzza S, Natella F, Unfer V, Sambuy Y, Monastra G. Enhancement of D-chiro-inositol transport across intestinal cells by alpha-Lactalbumin peptides. Eur Rev Med Pharmacol Sci. 2020 Oct;24(19):10143-10154. doi: 10.26355/eurrev_202010_23234. PMID 33090422
- [Background] Wang J, Aalaei K, Skibsted LH, Ahrne LM. Calcium bioaccessibility increased during gastrointestinal digestion of alpha-lactalbumin and beta-lactoglobulin. Food Res Int. 2023 Feb;164:112415. doi: 10.1016/j.foodres.2022.112415. Epub 2022 Dec 27. PMID 36737996
- [Background] Perego S, Del Favero E, De Luca P, Dal Piaz F, Fiorilli A, Cantu' L, Ferraretto A. Calcium bioaccessibility and uptake by human intestinal like cells following in vitro digestion of casein phosphopeptide-calcium aggregates. Food Funct. 2015 Jun;6(6):1796-807. doi: 10.1039/c4fo00672k. PMID 25927875
- [Background] Permyakov EA. alpha-Lactalbumin, Amazing Calcium-Binding Protein. Biomolecules. 2020 Aug 20;10(9):1210. doi: 10.3390/biom10091210. PMID 32825311
- [Background] Hirao M, Hashimoto J, Ando W, Ono T, Yoshikawa H. Response of serum carboxylated and undercarboxylated osteocalcin to alendronate monotherapy and combined therapy with vitamin K2 in postmenopausal women. J Bone Miner Metab. 2008;26(3):260-4. doi: 10.1007/s00774-007-0823-3. Epub 2008 May 11. PMID 18470667
- [Background] Kasukawa Y, Miyakoshi N, Ebina T, Aizawa T, Hongo M, Nozaka K, Ishikawa Y, Saito H, Chida S, Shimada Y. Effects of risedronate alone or combined with vitamin K2 on serum undercarboxylated osteocalcin and osteocalcin levels in postmenopausal osteoporosis. J Bone Miner Metab. 2014 May;32(3):290-7. doi: 10.1007/s00774-013-0490-5. Epub 2013 Jul 12. PMID 23846118
- [Background] Aaseth JO, Finnes TE, Askim M, Alexander J. The Importance of Vitamin K and the Combination of Vitamins K and D for Calcium Metabolism and Bone Health: A Review. Nutrients. 2024 Jul 25;16(15):2420. doi: 10.3390/nu16152420. PMID 39125301
- [Background] Defeudis G, Cardinali L, Eftekhariranjbar S, Massari MC, Migliaccio S. Male osteoporosis: the impact of lifestyle, from nutrition to physical activity. J Endocrinol Invest. 2025 May;48(5):1075-1083. doi: 10.1007/s40618-024-02517-w. Epub 2024 Dec 16. PMID 39680363